CLINICAL TRIAL: NCT06210256
Title: A Comparison of Unidirectional Valve Apparatus With Occluding the Non-ventilated Endobronchial Lumen for Lung Collapse During Video-associated Thoracoscopy: a Prospective Randomized Controlled Trial.
Brief Title: Compared Unidirectional Valve Apparatus and Occluding the Non-ventilated Endobronchial Lumen for Lung Collapse.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Peng Liang，MD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023HXFH012
Record Dates: First submitted 2024-01-04; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Video-assisted Thoracoscopic Surgery; One-Lung Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To guarantee the blinding of the surgeons and data recorders, a cover was placed over the patient's head and the DLT connector during the surgical operation. An independent investigator, who blinded to treatment assignment, carried out the postoperative assessment of lung collapse quality and subsequent follow-up visits. The anesthesiologist, who performed the DLT intubation, was the only study personnel unblinded to the randomization scheme and was not involved in data collection and analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the unidirectional valve group (Experimental): In the unidirectional valve group, as soon as disinfection and draping began, the lumen of the Y-connector to the non-ventilated lung was clamped and the unidirectional valve device was fastened to the bronchoscope port of the tracheal lumen to initial the one-lung ventilation.
  Interventions: Procedure: unidirectional valve apparatus
- the closed lumen group (Active Comparator): In the closed lumen group, as soon as disinfection and draping began, the lumen of the Y-connector to the non-ventilated lung was clamped, and the bronchoscope port of the tracheal lumen was sealed off from the atmosphere until pleural opening. When the pleura opened, the bronchoscope port opened to the air for 30 seconds before closing once more until the one-lung ventilation was completed.
  Interventions: Procedure: occluding the non-ventilated endobronchial lumen

INTERVENTIONS:
Procedure: unidirectional valve apparatus — In the unidirectional valve group, we attached the unidirectional valve device to the lumen's distal port when one-lung ventilation initiated.
  Arms: the unidirectional valve group
Procedure: occluding the non-ventilated endobronchial lumen — In the closed operative lumen group, we closed the lumen's distal port of non-ventilated lung when one-lung ventilation initiated.
  Arms: the closed lumen group

SUMMARY:
With the rapid advancement of thoracoscopic surgery in recent years, surgeons have set higher standards for the quality of non-ventilated lung collapse. In a prior investigation, we examined a unidirectional valve device that let air exit the non-ventilated side of the lung but not enter during ventilation and showed the use of this device during one-lung ventilation (OLV) for patients undergoing thoracoscopic surgery could speed up lung collapse, lower endogenous positive end-expiratory pressure, and have no discernible effects on oxygenation. In light of this, we conducted this study to further demonstrate, by comparison with the commonly used clinical technique of occluding the non-ventilated endobronchial lumen during one-lung ventilation, that this unidirectional valve device can quicken and enhance the quality of lung collapse without raising the risk of adverse events when used in thoracoscopic surgery.

DETAILED DESCRIPTION:
In this study, patients who meet the enrollment criteria will be randomized 1:1 to the unidirectional valve group or the closed lumen group.

After patients entered the operating room, their heart rate, mean arterial pressure, electrocardiogram, and pulse oxygen saturation were monitored. The electrodes of a bispectral index (BIS) Vista monitor were placed on the patient's forehead. The mask for oxygen inhalation at 6 L/min was then applied. Anesthesia was induced with 2mg midazolam, 0.3ug/kg sufentanil, 2-3mg/kg propofol and 0.3mg/kg cisatracurium using ideal body weight. Patients were intubated using a video double-lumen endotracheal tube [Disposable sterile double-lumen tracheal intubation, Nortier] by a senior anesthesiologist. Following confirmation of the double-lumen tube (DLT) placement position, two-lung ventilation was started at a respiratory rate of 15 breaths per minute, with an inspiratory to expiratory (I: E) ratio of 1:2, tidal volume of 8 ml/kg, and an inspired oxygen fraction (FiO2) of 0.8. Remifentanil (0.05-0.3 ug/kg/min) and propofol (4-12 mg/kg/h) were continuously infused to maintain anesthesia while the levels of BIS fluctuated between 40 and 60. The DLT placement location was verified again as soon as the disinfection and draping process started, and one-lung ventilation was initiated. In this study, we used a disposable plastic membrane glove and chopped off the fingers to create a unidirectional valve device. Our prior clinical experiment showed that this device permits gas in the non-ventilated lung to exit during exhalation, while ambient air could not enter via the collapsed cut hole during inhalation. In the unidirectional valve group, as soon as disinfection and draping began, the lumen of the Y-connector to the non-ventilated lung was clamped and the unidirectional valve device was fastened to the bronchoscope port of the tracheal lumen to initial the one-lung ventilation. In the closed lumen group, as soon as disinfection and draping began, the lumen of the Y-connector to the non-ventilated lung was clamped, and the bronchoscope port of the tracheal lumen was sealed off from the atmosphere until pleural opening. When the pleura opened, the bronchoscope port opened to the air for 30 seconds before closing once more until the one-lung ventilation was completed. The tidal volume was adjusted to 6 ml/kg during OLV, and the respiratory rate was set to 15 breaths per minute with a I:E ratio of 1:2 and FiO2 of 0.8. Positive expiratory pressure was not applied in this trial. After pleural opening, the thoracoscopic surgery procedure was captured on video using an electronic equipment. The anesthesiologist, who was blind to the specific lung collapse technique, watched the recordings after surgery and used a visual analogue scale to assess the quality of lung collapse at various time points. Bronchial suction was employed to foster lung collapse of the non-ventilated lung if there was no collapse or partial collapse of the lung during the surgical procedure. The number and timing of bronchial suction should be documented in detail. After surgery, patients were transferred to the post-anesthesia care unit (PACU) for continued monitoring. Throughout their hospital stay, the patients were visited daily, and any postoperative pulmonary issues were recorded in time until the patients were released from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* American Society of Anesthesiologists (ASA) physical status I to III
* Patients scheduled to undergo video-associated thoracoscopic surgery requiring one-lung ventilation

Exclusion Criteria:

A - pre-operative

1. anticipated difficult intubation
2. New York Heart Association (NYHA) heart failure class III/IV
3. body mass index≥35kg/m2
4. patients with abnormal expiratory recoil [forced expiratory volume in 1s (FEV1) less than 70% of predicted values
5. chronic obstructive pulmonary disease (COPD) or severe asthma
6. prior thoracic surgery or radiotherapy
7. a history of pleural or interstitial disease

B - post-randomization

1. the discovery of pleural adhesions following pleural opening
2. a delay of more than 25 minutes between the onset of one-lung ventilation and chest opening
3. the duration between the onset of one-lung ventilation and chest opening less than 10 minutes
4. a switch to thoracotomy as the type of surgical procedure
5. he occurrence of significant adverse events during the operation, such as severe bleeding (more than 1500ml), fatal arrhythmia, respiratory arrest, or cardiac arrest

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
The time needed for satisfactory lung collapse | The first 24 hours after surgery
  The outcome was measured from the initial of one-lung ventilation after clamping the non-ventilated lumen of DLT to the time of satisfactory lung collapse, graded via video view, by an independent investigator who was blinded to the lung collapse technique using a verbal analogue scale (0 = no lung collapse; 10 = total lung collapse). A score of eight for satisfactory lung collapse meant that the lung tissue had essentially collapsed, the surgical field was clearly visible, and the surgeons could carry out routine procedures.

SECONDARY OUTCOMES:
The quality of lung collapse | The first 24 hours after surgery
  An independent investigator viewed the video and scored the quality of lung collapse upon entering the thoracic cavity, and at 5, 10, 15, and 20 min following pleural opening using a verbal rating scale from zero to ten (0 = no lung collapse; 10 = total lung collapse).
The need for bronchial suction | Up to the end of the thoracoscopic surgery
  If there was no collapse or just partial collapse of the lung during the surgical procedure and it hindered the surgical operation, bronchial suction was used to promote lung collapse of the non-ventilated lung.
The development of intraoperative hypoxemia | Up to the end of the thoracoscopic surgery
  The development of intraoperative hypoxemia was defined as a decrease in peripheral blood oxygen saturation (SpO2) below 90% during surgical procedure.
The incidence of postoperative pulmonary complications | During hospital stay, an expected average of one week
  The patients developed one or more of the following postoperative pulmonary complications during hospitalization: respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonitis.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No